CLINICAL TRIAL: NCT06815627
Title: A Prospective, Multicenter, Phase III Clinical Evaluation of the Safety and Efficacy of NH002 as a Contrast Agent in Subjects Undergoing Cardiac Echocardiography
Brief Title: Safety and Efficacy Evaluation of NH002 as a Contrast Agent in Subjects Undergoing Cardiac Echocardiography
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Trust Bio-sonics, Inc. (Industry)
Collaborators: CMIC ASIA-PACIFIC, PTE. LTD., TAIWAN BRANCH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NH002-LV-02
Record Dates: First submitted 2025-01-21; First posted 2025-02-07 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Diseases
Keywords: Echo; Echocardiogram; Cardiac ultrasound; suboptimal; contrast agent; enhancing agent; LVO; LVEBD
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NH002 (Experimental): Subjects will undergo an unenhanced ultrasound examination and a NH002 contrast-enhanced examination (following intravenous (IV) doses of NH002: 2.5 µl/kg) on the same day.
  Interventions: Drug: NH002 (Perflutren Lipid Microspheres) Injectable Suspension

INTERVENTIONS:
Drug: NH002 (Perflutren Lipid Microspheres) Injectable Suspension — NH002 is formulated as a microbubble injectable suspension for intravenous administration. NH002 requires an activation process prior to use.

SUMMARY:
This is a Phase 3, prospective, open-label, multicenter study to assess the efficacy of NH002-enhanced echocardiography in subjects with suboptimal echocardiograms to opacify the left ventricular chamber and to improve the left ventricular endocardial border delineation compared with unenhanced echocardiography. The study also aims to investigate the safety and tolerability of NH002.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Ability to understand and the willingness to provide written informed consent
3. Having or suspected of having cardiac disease
4. Undergone a transthoracic echo within 30 days prior to NH002 dose administration, resulting in suboptimal LVEBD, as defined by 2 or more segments of 6 segments of the ventricular border that cannot be visualized reliably in any of the standard apical 4-, 2-, and 3-chamber views during the resting non-contrast ultrasound examination

Exclusion Criteria:

Subjects will be excluded from the study if one or more of the following exclusion criteria are applicable:

1. Any evidence of other severe or unstable cardiopulmonary and/or systemic hemodynamic conditions deemed unsuitable for the study by the investigator(s) prior to NH002 dose administration, including, but not limited to:

   1. ongoing or recent acute coronary syndrome within 6 months.
   2. uncontrolled serious ventricular arrhythmias.
   3. decompensated or inadequately controlled congestive heart failure (New York Heart Association Class IV).
   4. atrial fibrillation or current uncontrolled cardiac arrhythmias causing symptoms or hemodynamic compromise.
   5. uncontrolled hypertension (i.e., resting systolic blood pressure >200 mmHg or diastolic blood pressure >110 mmHg or arterial hypotension [defined as systolic blood pressure ≤ 90 mmHg]).
   6. acute aortic dissection.
2. Known or suspected hypersensitivity to one or more of the ingredients of NH002, perflutren, Definity®, or other echocardiographic contrast agents
3. Known or suspected hypersensitivity to polyethylene glycol, prior reactions to common polyethylene glycol-containing products such as colonoscopy bowel preparations, and certain laxatives (e.g., Miralax)
4. Received an investigational compound within 30 days before enrolling in the study
5. Received any contrast agent either intravascularly or orally within 48 hours prior to NH002 dose administration
6. Pregnant or lactating female. Exclude the possibility of pregnancy:

   1. testing on-site at the institution (serum or urine β-human chorionic gonadotropin) within 24 hours prior to the start of NH002 dose administration, and
   2. history of using an adequate and medically approved method of contraception to avoid pregnancy for at least 1 month prior to NH002 dose administration and willing to continue using the same method for the duration of the study, or
   3. surgical history (e.g., tubal ligation or hysterectomy), or
   4. postmenopausal with a minimum of 1 year without menses.
7. Serious medical or psychiatric illness/condition likely, in the judgment of the investigator, to interfere with compliance to protocol treatment/research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Endocardial Border Delineation (LVEBD) | Image data obtained pre-injection and within 10 minutes post-injection
  The first primary efficacy endpoint will be the change from baseline in total LVEBD scores (UEUS vs CEUS) defined using a 16-segment model derived from the standard 17-segment model, as assessed through blinded central reading. The LV endocardium of the standard apical 4-, 2-, and 3-chamber views is divided into 6 segments, with 2 basal, mid-, and apical segments in each view, of which 2 segments are shared in the standard apical 4- and 3-chamber views (i.e., a total of 16 segments in the 3 views). The 17th segment at the apex will not be scored since it does not connect to any part of the LV endocardial border. For each segment, LVEBD is graded as follows: 0 = inadequate border (border not visible); 1 = sufficient (border barely visible); 2 = good (border clearly visible). A total delineation score (0 to 32) is obtained by adding the scores from a total of the 16 segments in the 3 views.
Left Ventricular Opacification (LVO) | Image data obtained pre-injection and within 10 minutes post-injection
  The co-primary endpoint will be the proportion of subjects with adequate LVO defined by an LVO grade of +2 (moderate) or +3 (complete), as assessed through blinded central reading.

SECONDARY OUTCOMES:
The number and percentage of subjects with suboptimal echocardiography converted into optimal echocardiography | Image data obtained pre-injection and within 10 minutes post-injection
  Objective evaluation of the number and percentage of subjects with suboptimal echocardiography (based on the definition of inadequate LVEBD; i.e., at least two segments [combined chamber view] with an LVEBD score of 0) converted into optimal echocardiography following administration of study drug will be summarized for each reader.
Standard 12-lead ECG QT interval | From pre-injection to 24 hours post injection
  Standard 12-lead ECG QT interval assessed prior to injection and at 10 and 30 minutes after the end of injection; and at 24 hours after the end of injection
Blood Pressure (BP) | From pre-injection to 24 hours post injection
  Changes in BP assessed prior to injection and at 5, 10, and 30 minutes the end of after injection; and at 24 hours after the end of injection
Heart Rate (HR) | From pre-injection to 24 hours post injection
  Changes in HR assessed prior to injection and at 5, 10, and 30 minutes the end of after injection; and at 24 hours after the end of injection
SpO2 | From pre-injection to 24 hours post injection
  SpO2 assessed by pulse oximetry prior to injection and at 5, 10, and 30 minutes after the end of injection; and at 24 hours after the end of injection

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chung Yu, Principal Investigator — Taipei Veterans General Hospital, Taiwan; Chung-Lieh Hung, Principal Investigator — Mackay Memorial Hospital; Chih-Hui Chin, Principal Investigator — Cathay General Hospital; Hsin-Yueh Liang, Principal Investigator — China Medical University Hospital; Ning-I Yang, Principal Investigator — Chang Gung Memorial Hospital; Chien-Boon Jong, Principal Investigator — National Taiwan University Hospital Hsin-Chu Branch
Locations (6):
- Taiwan (6):
  - Keelung Chang Gung Memorial Hospital & Lovers Lake Branch, Keelung
  - China Medical University Hospital, Taichung
  - MacKay Memorial Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital Hsin-Chu Branch, Zhubei

IPD SHARING:
Plan to Share IPD: No